CLINICAL TRIAL: NCT02324699
Title: Corticosteroids as Co-Induction Agents With Vedolizumab in Crohn's Disease: a Double-blind Placebo Controlled Randomized Trial
Brief Title: Corticosteroids With Vedolizumab in Crohn's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Bruce E. Sands, Professor of Medicine Division of Gastroenterology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 14-2209
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
Keywords: Vedolizumab; Corticosteroids; Prednisone; Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Prednisone; Adrenal Cortex Hormones; vedolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone co-inductive therapy (Experimental): Prednisone 40 mg/day starting at week 0 for 2 weeks, tapered by 10 mg weekly to achieve 0 mg by end of week 5
  Interventions: Drug: Prednisone; Drug: Vedolizumab
- Placebo (Placebo Comparator): Identical placebo taper
  Interventions: Drug: Placebo; Drug: Vedolizumab

INTERVENTIONS:
Drug: Prednisone
  Other Names: corticosteroids
  Arms: Prednisone co-inductive therapy
Drug: Placebo
  Arms: Placebo
Drug: Vedolizumab — 300mg IV over 30 minutes. Both arms will receive vedolizumab at weeks 0, 2, and 6.
  Other Names: Entyvio

SUMMARY:
Use of co-induction with corticosteroid therapies may accelerate the remission rate when used with vedolizumab. Further, this may lead to higher rates of response and remission at week 10 than would be seen with vedolizumab monotherapy.

DETAILED DESCRIPTION:
This study will examine prednisone co-induction with vedolizumab in patients with Crohn's disease. To address questions regarding the effect of co-induction on mucosal healing, the study will include colonoscopic assessment of mucosal healing. Finally, colonic biopsies in this study will allow to elucidate further the mechanism of action of vedolizumab in Crohn's disease through immune phenotyping studies.

ELIGIBILITY:
Inclusion Criteria:

* Age at entry 18 to 70
* CDAI score > 220
* Concomitant azathioprine, methotrexate, or mercaptopurine permitted if dose has been stable for > 8 weeks. Prior anti-TNFα antibody use permitted but must be discontinued (>2 weeks from last dose) prior to initiation of vedolizumab.
* Documented ulceration on colonoscopy done at screening of 3 or more large ulcers or 10 or more aphthous ulcers
* Able to provide written informed consent.
* Patient is planned for or eligible to initiate vedolizumab

Exclusion Criteria:

* Concurrent use of anti-TNFα antibodies.
* No corticosteroids within prior 3 months (other than budesonide controlled ileal release)
* No stoma at the time of enrollment
* No absolute contraindication to systemic corticosteroid use such as hypersensitivity to any part of the formulation, systemic fungal infection, or recent administration of live or live attenuated vaccine within prior two weeks.
* Pregnant women or plans for pregnancy within 3 months of study inclusion
* Presence of stoma, more than three small-bowel resections, or documented history of short bowel syndrome
* Intestinal stricture requiring surgery
* Abdominal abscess
* Inability or unwillingness to provide informed consent
* Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04; Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce E Sands, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai Hospital
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened in August 2015,and one participant enrolled almost a year later.
Pre-assignment Details: Study is double blind and unknown which arm participant was randomized into. Study was never unblinded.
Groups:
- Prednisone Co-inductive Therapy: Prednisone vs Identical placebo taper
  Prednisone 40 mg/day starting at week 0 for 2 weeks, tapered by 10 mg weekly to achieve 0 mg by end of week 5
  Vedolizumab: 300mg IV over 30 minutes. Both arms will receive vedolizumab at weeks 0, 2, and 6.
Period: Overall Study
Arm/Group | Prednisone Co-inductive Therapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — study terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Prednisone Co-inductive Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Crohn's Disease Activity Index (CDAI)
Description: Clinical remission, defined as CDAI < 150, in group with steroid co-induction vs. placebo co-induction. The purpose of this crohn's disease activity index (CDAI) calculator is to gauge the progress or lack of progress for people with crohn's disease. CDAI scores below 150 indicate a better prognosis than higher scores
Time Frame: baseline, week 6, week 10
Measure: Number; unit: score on a scale
Arm/Group | Prednisone Co-inductive Therapy
Number analyzed (Participants) | 1
score on a scale
  Baseline | 263
  Week 6 | 112.6
  Week 10 | 137.5

2. Secondary Outcome: Change in Simple Endoscopic Score for Crohn's Disease (SES-CD)
Description: The SES-CD tool is used to quantify and compare inflammatory load. The Simple Endoscopic Score for Crohn Disease (SES-CD) assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence of stenosis. Each item is scored from 0-3, with total score from 0-60. Higher score indicates more severe endoscopic activity.
Time Frame: baseline and week 10
Measure: Number; unit: score on a scale
Arm/Group | Prednisone Co-inductive Therapy
Number analyzed (Participants) | 1
score on a scale
  Baseline | 24
  Week 10 | 18

3. Secondary Outcome: Change in C-Reactive Protein (CRP)
Description: Comparison of absolute change in CRP from baseline to week 10. C-reactive protein is produced by the liver. The level of CRP rises when there is inflammation throughout the body.
Time Frame: baseline and week 10
Measure: Number; unit: mg/L
Arm/Group | Prednisone Co-inductive Therapy
Number analyzed (Participants) | 1
mg/L
  baseline | 11.0
  week 10 | 43.0

4. Secondary Outcome: Change in Calprotectin
Description: Comparison of absolute change in calprotectin from baseline to week 6. Calprotectin is a stool (fecal) test that is used to detect inflammation in the intestines.
Time Frame: baseline, week 6 and week 10
Population: data not collected
Arm/Group | Prednisone Co-inductive Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Prednisone Co-inductive Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study terminated due to enrollment difficulty.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT02324699/Prot_SAP_000.pdf